CLINICAL TRIAL: NCT06137599
Title: GCS Survey: "GHB IN CHEMICAL SUBMISSION: MYTH OR REALITY?"
Acronym: GCS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Mission Interministérielle de Lutte contre les Drogues et les Conduites Addictives - MILDECA (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP230579
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: CHEMICAL SUBMISSION
Keywords: CHEMICAL SUBMISSION; Chemical vulnerability; Drug facilitated Crime; Gamma hydroxybutyrate; Capillary analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — capillary sampling and analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Capillary analysis — Samples taken between 2 and 6 months after the presumed events. A pre-analytical treatment of the hair (washing, fragmentation), followed by detection by high-resolution mass spectrometry is carried out by an expert laboratory to search for both GHB and psychoactive drugs.

SUMMARY:
According to the media, GHB is the main substance used for chemical submission. The national survey conducted by the Addictovigilance centre of Paris on drug-facilitated assaults shows that GHB is used, but only in a very small proportion of cases. However, the short detection times for this substance point to its possible under-detection (06-09h in blood, 10-12h in urine). A pilot research protocol in Ile de France focusing on capillary analysis is therefore being proposed to volunteer victims to overcome this bias and answer this question: is the massive use of GHB in chemical submission a myth or a reality?

DETAILED DESCRIPTION:
The Addictovigilance center of Paris (CEIP-A) has been responsible for the national chemical submission survey under the supervision of the French National Agency for the Safety of Medicines and Health Products (ANSM) since 2003, using data from expert toxicology laboratories, forensic police and forensic medicine departments. With 20 years' experience in the criminal use of substances, the center draws up an annual report on substance-facilitated assaults in order to put in place appropriate, up-to-date prevention measures.

In 2021, the #balancetonbar movement emerged in Brussels and spread like a shockwave across Belgian cities and Europe. On Instagram, women spoke out about the extent of drug-facilitated sexual assault (DFSA) in nightclubs and denounced the " laissez faire " attitude of the political authorities. The movement is resonating in France and getting louder : #balancetonbar has now been joined by #MetooGHB, which puts the so-called "rape drug" in the spotlight. But what's really going on?

A retrospective study of the national survey data from 2010 to 2019 reports only 26 chemical submissions (CS) attributable to GHB/GBL out of 617 CS identified (4.2%) among 4349 suspected cases. However, this study highlights all the limits to the disclosure of GHB (low proportion of complaints filed, speed of elimination of this substance from the usual matrices, insufficient number of court orders for hair analysis).

With the aim to eliminate the limitations identified as far as possible and answer the question "Is the massive use of GHB in chemical submission a myth or a reality?", a pilot research protocol, centred on capillary analysis, is being proposed to 200 victims in the Ile de France region.

This is a non-interventional, multi-centre, category 3 study, the only acts (hair sampling) or procedures (chemical submission declaration form) are risk-free and do not affect the management of participants.

Victims are included whether or not they have lodged a complaint, in collaboration with forensic medicine departments, HIV and STI screening Center and Victim Support Associations. Referred to the parisien CEIP-A, 3 strands of hair are sampled after an interview in which the victim's history and voluntary drug use data were taken. A pre-analytical treatment of the hair (washing, fragmentation), followed by detection by high-resolution mass spectrometry is carried out by an expert laboratory in search of GHB and other known chemical submission agents (illicit drugs and psychoactive medicines).

To meet our objective, a comparative study of the results of the GCS protocol and the survey history was carried out using an exact binomial test. This study will also provide an opportunity for a more general discussion of the value of hair analysis in the detection of chemical submission agents.

ELIGIBILITY:
Inclusion Criteria:

* Victims over the age of majority (≥ 18 years) on the day of the alleged events
* With a medical history leading to the suspicion of chemical submission:
* Presence of evocative clinical signs (amnesia and/or behavioural disorders and/or neurological disorders and/or other somatic disorders, etc.) AND
* In the presence of potential criminal acts (suspected or proven assault or attempted assault).
* French speaking
* Having been informed of the search

Exclusion Criteria:

* - Victims who were minors (<18 years) on the day of the alleged events.
* Victims who usually use GHB/GBL recreationally.
* Suspecting administration of a harmful substance with no crime or offence committed at the time and no attempted assault
* Victims of needle spiking
* Victims with very short hair (<3 cm), bald or shaven heads
* Victims who have exceeded the maximum time limit for taking a hair sample (6 months after the event)
* Do not speak French
* Oppose to participating in the study
* Victims presenting a psychotic or cognitive syndrome likely to impair judgement Victims placed under guardianship or legal protection (article L11-22-2 CSP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any person suspecting of having been the victim of chemical submission (attack after taking a substance without the victims' knowledge or under threat
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-03-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Evidence of exogenous GHB intake without the knowledge of the victims through hair analysis. | Samples taken between 2 and 6 months after the presumed events: GHB analysis in the hair can no longer be interpreted after 6 months due to the hydrosoluble nature of GHB and repetitive hair washing.
  A double CEIP-A/Expert Laboratory interpretation is carried out according to the evaluation criteria defined by the national chemical submission survey Steering Committee.

SECONDARY OUTCOMES:
Evidence of the use of a psychoactive substance (other than GHB) without the knowledge of the victims via capillary analysis. | Samples taken between 2 and 6 months after the presumed events.
  A double CEIP-A/Expert Laboratory interpretation is carried out according to the evaluation criteria defined by the national chemical submission survey Steering Committee.

CONTACTS AND LOCATIONS:
Overall Officials: Leïla CHAOUACHI, PharmD, Study Chair — APHP(ASSISTANCE PUBLIQUE DES HOPITAUX DE PARIS; Anne Batisse, PharmD, Study Director — APHP(ASSISTANCE PUBLIQUE DES HOPITAUX DE PARIS
Locations (3):
- France (3):
  - Laetitia LASNE, Bondy
  - Elisabeth ALCARAZ, Paris
  - Leila CHAOUACHI, Paris

IPD SHARING:
Plan to Share IPD: No